CLINICAL TRIAL: NCT05701085
Title: Prospective Cohort Study of a Patient Navigator PRE-ACT Educational Intervention to Promote Decision Making About Clinical Trials Among Racial and Ethnic Minorities
Brief Title: Patient Navigator PRE-ACT Educational Intervention to Promote Decision Making Among Minorities
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE3522
Record Dates: First submitted 2022-11-29; First posted 2023-01-27 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Educational Intervention; Minorities
Keywords: PRE-ACT
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRE-ACT Adaptation (Experimental): At the scheduled oncologic visit: consent obtained and all participants will complete the Demographics/Clinical Characteristics survey and Pre-Intervention Survey
  Within 3 months of consent: tailored educational intervention and patient navigation program will take place and the scored Pre-Intervention survey will be used to generate a list of barrier for each patient. The patient will be asked to view educational videos on an iPad that correspond with each identified barrier. Afterwards, the patient navigator will lead a discussion based on the topics discussed.
  Within 4 weeks of the educational video: the participant will be contacted via phone to complete a Post-Intervention Survey that assesses knowledge, attitudes, and preparation related to participation in clinical trials
  Two years after intervention: chart review will be performed to assess if the patient participated in a clinical trial.
  Interventions: Other: Educational Intervention

INTERVENTIONS:
Other: Educational Intervention — The intervention will occur at a separate dedicated in-person visit with the patient navigator estimated to last 30-45 minutes. The Pre-Intervention Survey will be scored to generate a list of barriers identified for each patient. This list of barriers will be reviewed by the patient navigator prior to the intervention date. The patient will be asked to view educational videos on an iPad that correspond with each identified barrier. Afterwards, the patient navigator will lead a discussion based on the topics discussed.

SUMMARY:
This study focuses on psychosocial barriers at the patient level with the goal of promoting high quality decision making around clinical trials participation. The proposed study adapts the PRE-ACT model to racial and ethnic minority patients who were underrepresented in the original PRE-ACT study and will be combined with a patient navigator model.

DETAILED DESCRIPTION:
The primary objective of the proposed research is to employ a non-directive method to improve preparedness for consideration of clinical trials among racial minority patients by providing tailored information to address knowledge and attitudes towards clinical trials. This model has been previously studied in a primarily white, well-educated population. It is unknown how well this model adapts to meet the needs of diverse patient populations.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a diagnosis of either advanced (metastatic) cancer or early stage disease for which they are undergoing oncological work-up, treatment or surveillance
* Participants must be at least 18 years of age
* Participants have a non-white race or Hispanic ethnicity recorded in their patient demographics in the electronic medical record
* Participant must have a life expectancy greater than three months based on the primary oncology team's clinical assessment.
* Participants must be able to read and verbally communicate in English.
* Participants must provide written informed consent.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-04-24 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in knowledge regarding cancer clinical trials after the intervention | Up to 4 months
  Change in knowledge regarding cancer clinical trials after the intervention will be assessed by change in Pre and Post Intervention Survey Knowledge Score (scored from Items 1-8) with a higher score correlating to a greater change in knowledge.
Change in attitudes regarding cancer clinical trials after the intervention | Up to 4 months
  A change in attitude will be recorded using changes in Pre and Post Intervention Survey Attitude Scores (scored from Items 9-21) with a higher score correlating to a greater change in attitude.

OTHER OUTCOMES:
Rate of racial/ethnic minority participation in cancer clinical trials before and after the intervention (exploratory outcome) | Up tp 28 months
  Number

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Chiec, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States